CLINICAL TRIAL: NCT02501395
Title: MRI in Patients With Kennedy Disease
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Julia Dahlqvist, MD, MD, Rigshospitalet, Denmark
Other Study IDs: H-15006316
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Bulbo-Spinal Atrophy, X-Linked; Kennedy Disease
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patients with Kennedy disease: Men over 18 years old with confirmed Kennedy disease.
  Interventions: Other: No intervention, observational
- Healthy, voluntary controls: Gender and age matched healthy, voluntary controls.
  Interventions: Other: No intervention, observational

INTERVENTIONS:
Other: No intervention, observational

SUMMARY:
Kennedy disease is an inherited neuromuscular disorder that is characterized by progressive muscle wasting and weakness. It typically starts with muscle spasms and tremors in the arms, followed by muscle weakness and atrophy of muscles in the arms and legs. The facial and bulbar muscles are also involved. However, the muscle involvement pattern has not been investigated systemically in Kennedy disease.

The primary aim of the study is to investigate the muscle involvement in patients with Kennedy disease using MRI. Secondary aims are to examine disease severity and to test MRI as a potential outcome measure for future clinical trials in Kennedy disease.

Approximately 40 patients with Kennedy disease and 20 gender and age matched healthy voluntary controls will be recruited. The study consists of one visit per subject lasting 4-5 hours.

ELIGIBILITY:
Patients with Kennedy disease:

Inclusion Criteria:

* Confirmed Kennedy disease

Exclusion Criteria:

* All contraindications for undergoing an MRI scan

Healthy controls

Inclusion Criteria:

* Fit age and gender criteria

Exclusion Criteria:

* All contraindications for undergoing an MRI scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons in Denmark diagnosed with Kennedy disease is invited to the study.
  Gender and age matched controls will be recruited to a control group.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Muscle fat fraction | One MRI scan per subject (exam lasts approximately 60 min.)
  The Dixon MRI will be used to quantify the fat fraction in skeletal muscle.

SECONDARY OUTCOMES:
Muscle strength | One muscle strength test per subject (exam lasts approximately 60 min.)
  Isokinetic muscle dynamometry will be used to measure muscle strength.
Minimal dataset for data collection in Kennedy disease | Data will be collected once for patients with Kennedy disease (exam lasts approximately 90 min.)
  The 'minimal dataset for data collection in Kennedy disease' will be used to investigate the clinical spectrum of Kennedy disease.

CONTACTS AND LOCATIONS:
Overall Officials: Julia R Dahlqvist, MD, Principal Investigator — Copenhagen Neuromuscular Center, Department of Neurology, Rigshospitalet, Copenhagen University
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

REFERENCES:
- See also: The homepage of Copenhagen Neuromuscular Center, Denmark. — http://neuromuscular.dk